CLINICAL TRIAL: NCT05074602
Title: A Randomized, Double-Blind, Double-Dummy, Parallel Fluconazole Controlled, Multicenter Phase III Clinical Study to Evaluate the Efficacy and Safety of SHR8008 vs. Fluconazole in Subjects With Recurrent Vulvovaginal Candidiasis (RVVC)
Brief Title: A Study to Evaluate the Efficacy and Safety of SHR8008 vs. Fluconazole in Subjects With Recurrent Vulvovaginal Candidiasis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR8008-301
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Recurrent Vulvovaginal Candidiasis
MeSH Terms: conditions — Candidiasis, Vulvovaginal | interventions — Fluconazole

STUDY DESIGN:
Intervention Model Description: A Randomized, Double-Blind, active controlled, parallel groups, Multicenter Phase III Clinical Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR8008 (Experimental)
  Interventions: Drug: SHR8008
- Fluconazole (Active Comparator)
  Interventions: Drug: Fluconazole

INTERVENTIONS:
Drug: SHR8008 — Dosing frequency: During Part 1, administered orally once daily for 2 days. During Part 2, administered orally once weekly for 11 weeks starting from Week 3, Route of administration: oral
  Arms: SHR8008
Drug: Fluconazole — Dosing frequency: During Part 1, administered orally 3 sequential doses (every 72 hours), During Part 2, administered orally once weekly for 6 Months starting from Week 3. Route of administration: oral
  Arms: Fluconazole

SUMMARY:
The purpose of this study is to evaluate the Efficacy and Safety of SHR8008 capsule In Subjects With Recurrent Vulvovaginal Candidiasis

ELIGIBILITY:
Inclusion Criteria:

1. Females, ≥18 and ≤75 years old.
2. Have a history of RVVC at screening.
3. Suitable for oral therapy and able to swallow capsules intact.
4. Subjects of childbearing potential must use highly effective contraceptive measures throughout the study.
5. Willing to sign the informed consent form to participate in this study.

Exclusion Criteria:

1. Presence of concomitant vulvovaginitis caused by other pathogens.
2. Have a history of cervical cancer, or "cervical intraepithelial neoplasia or malignancy" or "atypical squamous cells of undetermined significance (ASCUS)" as indicated by Pap test or other tests reported within 1 year before screening (not applicable to subjects with a history of total hysterectomy).
3. Any condition that, in the opinion of the investigator, could impact drug absorption, distribution, or elimination.
4. Moderate to severe hepatic and/or renal disorders.
5. Significant laboratory abnormality at screening.
6. QTc interval greater than 470 ms or other clinically significant ECG abnormality at screening.
7. Have received systemic or vulvovaginal antifungal drugs, antibacterials, antitrichomonal, CYP3A4 substrates or inducers or inhibitors, and vulvovaginal corticosteroids within 7 days prior to randomization.
8. Have received any estrogen replacement therapy or vaginal topical products.
9. Have received systemic corticosteroid therapy within 30 days or systemic immunosuppressant therapy within 90 days prior to randomization;
10. Have planned surgery or other medical procedures that may impact compliance with the protocol;
11. Known history of hypersensitivity or intolerance to azole antifungal drugs.
12. History of narcotic or drug abuse or alcoholism, or any other medical, psychiatric or social condition that in the investigator's opinion could preclude compliance with the protocol.
13. Women who are pregnant or lactating, or planning to become pregnant during the study period.
14. Have received VT-1161 study medication in a previous study or received any investigational medicinal product (IMP) in a clinical study within 5 half-lives of that IMP prior to screening (if the half-life is unknown, 60 days prior to screening);
15. other conditions unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with one or more culture-verified VVC episodes during the study. | 50 weeks

SECONDARY OUTCOMES:
The proportion of subjects with resolved VVC episode (clinical signs and symptoms score of < 3) during induction phase | Day 14
The proportion of subjects with 2 culture-verified VVC episodes during the study. | week 50
The proportion of subjects with ≥ 3 culture-verified VVC episodes during the study. | week 50
The proportion of subjects with one or more culture-verified VVC episodes during the maintenance phase and follow-up phase. | Week 3 through Week 50
Time to first recurrence of a culture-verified VVC episode during the maintenance phase and follow-up phase. | Week 3 through Week 50
The proportion of subjects with at least one positive culture for Candida species during the maintenance phase and follow-up phase | Week 3 through Week 50
The proportion of subjects receiving rescue treatment during the maintenance phase and follow-up phase. | Week 3 through Week 50
The proportion of subjects with clinical cure (defined as the absence of all signs and symptoms of VVC) at the end of induction phase . | Day 14
The proportion of subjects with mycological cure (defined as vaginal swab culture negative for growth of Candida species) at the end of induction phase. | Day 14
The proportion of subjects with therapeutic cure (clinical cure plus mycological cure) at the end of induction phase. | Day 14
The proportion of subjects with therapeutic cure, clinical cure, and mycological cure during the maintenance phase. | Day 14
The proportion of subjects with one or more culture-verified VVC episode during the maintenance phase | Week 3 through Week 13
The proportion of subjects with at least one positive culture for Candida species during the maintenance phase | Week 3 through Week 13
The proportion of subjects with one or more culture-verified VVC episode during the maintenance phase | Week 3 through Week 26
The proportion of subjects with at least one positive culture for Candida species during the maintenance phase | Week 3 through Week 26
The proportion of subjects with one or more culture-verified VVC episodes during the follow-up phase. | Week 27 through Week 50
The proportion of subjects with at least one positive culture for Candida species during the follow-up phase | Week 27 through Week 50

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided